CLINICAL TRIAL: NCT01694303
Title: Computerized Interventions for College Students' Cognitive Functioning and Mental Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amit Etkin, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-24519
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Engaging computerized tasks (Active Comparator): Participants will log into a personalized website and engage in computerized tasks online.
  Interventions: Behavioral: Computerized Neurobehavioral Intervention
- Neurobehavioral computerized tasks (Experimental): Participants will log into a personalized website and engage in computerized tasks online.
  Interventions: Behavioral: Computerized Neurobehavioral Intervention

INTERVENTIONS:
Behavioral: Computerized Neurobehavioral Intervention — Targeted, computerized interventions completed from the participants' own home on a computer.

SUMMARY:
The present study will explore the effectiveness of a computer based neurobehavioral intervention in improving cognition and emotion regulation in a college freshmen population. It will increase understanding of emotion-regulation and cognition at a neural-circuit level and aid development of new interventions for emotion regulatory problems.

ELIGIBILITY:
Inclusion Criteria:

* internet access

Exclusion Criteria:

* lifetime psychotic disorder,
* past-year substance dependence

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Emotion-regulation - behavioral and fMRI | 3-month

SECONDARY OUTCOMES:
Cognition - executive function behavioral reaction time | 3-month

CONTACTS AND LOCATIONS:
Overall Officials: Anett Gyurak, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Department of Psychiatry and Behavioral Sciences, Stanford, California, United States

REFERENCES:
- [Derived] Gyurak A, Patenaude B, Korgaonkar MS, Grieve SM, Williams LM, Etkin A. Frontoparietal Activation During Response Inhibition Predicts Remission to Antidepressants in Patients With Major Depression. Biol Psychiatry. 2016 Feb 15;79(4):274-81. doi: 10.1016/j.biopsych.2015.02.037. Epub 2015 Mar 27. PMID 25891220